CLINICAL TRIAL: NCT03976414
Title: Reach and Teach: Translating "Mind Over Matter: Healthy Bowels, Healthy Bladder" for Digital Delivery
Brief Title: Mind Over Matter: Electronic Bladder and Bowel Continence Self-management Program
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-1147; SMPH/OBSTET & GYNECOL/OBSTET & (Other: UW, Madison); A532800 (Other: UW, Madison)
Record Dates: First submitted 2019-05-06; First posted 2019-06-06 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2020-09

CONDITIONS: Incontinence, Urinary; Incontinence Bowel
MeSH Terms: conditions — Urinary Incontinence; Encopresis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- eMOM website users: Any woman who visits the "research" tab on the eMOM website will see an invitation to participate in a research study about the impact of the website on her bladder and bowel symptoms. Women may use the intervention (the website) regardless of whether they opt to participate in the research study.
  The intervention is the use of the website (eMOM), which is the electronic adaption of the program, Mind Over Matter: Healthy Bowels, Healthy Bladder (MOM), a small-group, community-based health promotion program that builds skills and self-efficacy to make behavior changes that improve urinary and bowel symptoms among older women with incontinence.
  Interventions: Other: eMOM

INTERVENTIONS:
Other: eMOM — The intervention is the use of the website (eMOM), which is the electronic adaption of the program, Mind Over Matter: Healthy Bowels, Healthy Bladder (MOM), a small-group, community-based health promotion program that builds skills and self-efficacy to make behavior changes that improve urinary and bowel symptoms among older women with incontinence.
  Other Names: Mind Over Matter: Healthy Bowels, Healthy Bladder" (MOM)

SUMMARY:
The objective of this study is to (1) use participatory ergonomics to adapt and in-person 3-session intervention: Mind Over Matter: Healthy Bowels, Healthy Bladder (MOM) to an electronic program (eMOM), and to (2) compare and characterize eMOM's reach when marketed via community agencies versus Facebook advertising and to collect qualitative and quantitative data about effectiveness and uptake of key behaviors using electronic surveys and phone interviews. The study will also collect information from community agencies that might implement eMOM about its perceived value and their willingness and capacity to implement such a program.

DETAILED DESCRIPTION:
More than half of patients hospitalized with serious illness rated urinary and bowel incontinence as a state worse than death in a 2016 JAMA (The Journal of the American Medical Association) internal medicine study - worse than relying on a breathing machine, being unable to get out of bed, or being confused all the time. Unfortunately, over 60% of community-dwelling women over age 65 suffer from urinary and/or bowel incontinence, accounting for a combined annual cost in excess of $30 billion. In addition to their impact on quality of life, social isolation, and depression, urinary and bowel incontinence increase caregiver burnout, risk for falls, hospitalization, and nursing home placement. However, despite the existence of effective treatments, over half of women with urinary incontinence and two-thirds of women with bowel incontinence do not seek medical care. Interventions to promote continence in healthcare settings thus reach fewer than half of those in need.

At University of Wisconsin, research team developed "Mind Over Matter: Healthy Bowels, Healthy Bladder" (MOM), which is a small-group, community-based health promotion program that builds skills and self-efficacy to make behavior changes that improve urinary and bowel symptoms among older women with incontinence. Delivered by a trained facilitator, MOM allows senior women to improve their symptoms without seeking medical care. In the randomized, controlled trial (RCT) including 122 women in 6 Wisconsin communities, more than 70% of participants (versus 23% of controls, p<.0001) achieved improvement in urinary incontinence and 55% (versus 26% of controls, p = .0015) achieved improvement in bowel incontinence three months following completion of the program, corresponding to a number-needed-to-treat of 3 for urinary incontinence improvement and 4 for bowel incontinence improvement.

However, community-based, in-person programs like MOM continue to suffer limited adoption, implementation, and reach. Many agencies that adopt and implement such health promotion programs are under-resourced and often staffed by volunteers. To ensure intervention fidelity, programs like MOM require a large commitment from their resource-stressed hosting agencies. Implemented using a "train the trainer" approach organized by the Wisconsin Institute for Healthy Aging (WIHA), MOM requires community facilitators to attend a 2-day training and then run the workshop series at least twice annually. In addition to the 2-day training, it requires approximately 24 person-hours to offer a single MOM workshop series. If the trained facilitator leaves or is redirected to other activities, the community agency can no longer implement or maintain the program without sending another staff member to be trained. In addition to these hurdles at the organization level, there are barriers at the individual level.

In a recent collaboration with the Survey of the Health of Wisconsin (SHOW), it was observed that fewer than 20% of women with incontinence (mean age 55 years old) reported being likely to attend a continence promotion program with the current, in-person MOM format. In qualitative interviews, women expressed concerns about the time commitment, caregiver responsibilities at home, issues related to travel (inclement weather, excessive distance to reach a community center), and privacy, given the sensitive nature of incontinence. In contrast, 65% of women with incontinence reported being likely to participate in an electronic continence promotion program, increasing potential reach three-fold.

Adaptation of the in-person MOM workshop to an electronic format (eMOM) has the potential to overcome both individual and organizational hurdles, maximizing reach and minimizing barriers to consistent implementation and maintenance. Women with incontinence can complete the modules in privacy, at their convenience, and at their own pace. In contrast to the commitment required for a community agency to implement the in-person MOM workshop, eMOM can be implemented using whatever strategies the agency uses to share other electronic resources with their members. eMOM can also be implemented via mass media, such as Facebook. Women age 65+ account for 11.6% of all Facebook users, and there are more than 200,000 monthly active users in this demographic in Wisconsin alone.

The proposed research will provide invaluable information about the feasibility and reach of implementing an electronic health promotion program through mass media versus through existing community agencies - information applicable not just to continence promotion but also to other health promotion programs trying to overcome similar barriers to reach, implementation, and maintenance.

ELIGIBILITY:
Inclusion Criteria:

* be able to access the eMOM website via internet
* must be able to speak and read English
* at least 18 years old
* female.

Exclusion Criteria:

* no access to internet
* no email address

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: While eMOM will be promoted specifically for older women, women of any age may access the program and participate in the study if they so choose.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Response on global perception of improvement (GPI) tool at 4 months | 4 months
  Global perception of improvement (GPI) is a tool for Global Rating of Patient Satisfaction and Perceptions of Improvement.
  Question asked: Overall, do you feel that you are? Response can be chosen from the options: Much Better, Better, About the same, Worse, Much worse

SECONDARY OUTCOMES:
Change in the response of Global patient satisfaction question (PSQ) | 1 month, 4 months, 6 months
  Patient satisfaction will be measured with the question: How satisfied are you with your progress in this program? (completely, some-what, not at all)
Change in patient estimated percent improvement (EPI) | 1 month, 4 months, 6 months
  For EPI, Patients will be asked to estimate how much better they were on a scale from 0% (no better) to 100%(completely better)
Change in response on global perception of improvement (GPI) at 1 month and 6 months | 1 month, 6 month
  Global perception of improvement (GPI) is a tool for Global Rating of Patient Satisfaction and Perceptions of Improvement.
  Question asked: Overall, do you feel that you are? Response can be chosen from the options: Much Better, Better, About the same, Worse, Much worse
Differences in scores of the International Consultation on Incontinence Questionnaire-Urinary Incontinence (ICIQ-UI) | Baseline, 1 month, 4 month, 6 month
  ICIQ-UI is a subjective measure of severity of urinary loss and quality of life for those with urinary incontinence. It is scored on a scale from 0-21. Based on the score participant can be placed in four severity categories: slight (1-5), moderate (6-12), severe (13-18) and very severe (19-21)
Differences in scores of the St. Mark's Incontinence Scale (aka Vaizey) | baseline, 1 month, 4 month, 6 month
  St. Mark's Incontinence Scale (aka Vaizey) will be used to assess the severity and the outcome of MOM intervention
  Never: no episodes in the past 4 weeks rarely: 1 episode in the past 4 weeks sometimes: > 1 episode in the past 4 weeks, but,1 a week; Weekly: 1 or more episodes a week but,1 a day Daily: 1 or more episodes a day
  Scores will be assigned for each row (Never=0, Rarely=1, Sometimes=2, Weekley=3, Daily=4 )
  Score will be added from each row. Cumulative minimum score=0 perfect continence; Cumulative maximum score will be 24= totally incontinence
Self-reported behavior changes: change in the frequency of pelvic floor muscle exercises | baseline, 1 month, 4 month, 6 month
  Frequency of pelvic floor muscle exercises
Self-reported behavior changes: change in fluid intake | baseline, 1 month, 4 month, 6 month
  Self-reported behavior changes: fluid intake
Self-reported behavior changes: change in fiber intake | baseline, 1 month, 4 month, 6 month
  Self-reported behavior changes: change in fiber intake
Self-reported coping changes: change in types of pad used | baseline, 1 month, 4 month, 6 month
  Self-reported coping changes: change in types of pad used
Self-reported coping changes: change in number of pads used | baseline, 1 month, 4 month, 6 month
  Self-reported coping changes: change in number of pads used
Self-reported changes: change in the money-spent on buying products to manage their incontinence | baseline, 1 month, 4 month, 6 month
  It will be measured by asking participants question that how much money have they spent on products (such as pads, undergarments, or plugs) to manage their bladder and/or bowel symptoms in the last month.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Brown, MD, Principal Investigator — UW-Madison Obstetrics and Gynecology
Locations (1):
- University of Wisconsin-Madison School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No